CLINICAL TRIAL: NCT05482503
Title: Clinical Investigation to Evaluate the Effectiveness and Safety of ECG App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huawei Device Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HWECG-001
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atrial Fibrillation (Experimental)
  Interventions: Device: 12-Lead ECG(I-lead)
- Premature beats (Experimental)
  Interventions: Device: 12-Lead ECG(I-lead)
- Sinus Rhythm (Experimental)
  Interventions: Device: 12-Lead ECG(I-lead)

INTERVENTIONS:
Device: 12-Lead ECG(I-lead) — All participants will simultaneously record 12-lead ECGs(I-lead)

SUMMARY:
The purpose of this study is to verify the effectiveness and safety of the Huawei Device software (ECG APP), which can be used to analyze, store and display the ECG data transmitted by the single-lead ECG acquisition device. The software can be used for the analysis of sinus rhythm, atrial fibrillation, and premature beats(ventricular premature beats and atrial premature beats) in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old, regardless of gender;
2. Participants who meet one of the following conditions according to the medical history in the past 3 months or the ECG during the screening period:

   1. Patients with normal sinus rhythm;
   2. Patients with persistent or permanent paroxysmal atrial fibrillation or in the onset of paroxysmal atrial fibrillation;
   3. Patients with frequent premature beats (more than 5 per minute) or in the onset of premature beats;
3. Patients who have good compliance, and can cooperate to complete this research by himself/herself; 4）Patients who volunteer to participate and have signed an informed consent form.

Exclusion Criteria:

1. Patients using cardiac pacemakers or implantable cardioverter defibrillators (ICD);
2. Patients with atrioventricular block or bundle branch block;
3. Patients with significant sinus arrhythmia, sinus arrest or sick sinus syndrome;
4. Patients with interpolated premature beats, junctional premature beats, or escape rhythms;
5. Patients with atrial tachycardia, atrial flutter, ventricular tachycardia, ventricular flutter, or ventricular fibrillation;
6. Patients with a resting heart rate of slower than 50 beats/minute or faster than 110 beats/minute;
7. Patients with atrial fibrillation complicated with premature beats;
8. Patients who are critically ill, making it difficult to make an accurate assessment of the effectiveness and safety of the device;
9. Patients who suffer from tremor diseases or chorea, making it difficult to complete the examination quietly;
10. Patients with bullous diseases or large-area skin rashes that are not suitable for body surface electrode recording;
11. Patients whose skin is allergic to ethanol;
12. Patients with contagious skin diseases;
13. Patients with a history of mental illness or with cognitive impairment;
14. Patients who have participated in other clinical investigations within the past 30 days that may affect this investigation; 15） Other conditions that the investigators consider inappropriate for participation in the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of atrial fibrillation identification | 30seconds
Sensitivity and specificity of premature beat identification | 30seconds
Sensitivity and specificity of sinus rhythm identification | 30seconds

SECONDARY OUTCOMES:
Detection rate of ventricular premature beats and atrial premature beats | 30seconds
Total coincidence rate of measurement and identification | 30seconds
ECG waveform similarity | 30seconds
R wave amplitude consistency | 30seconds
Heart rate accuracy | 30seconds
Software usability | 30seconds

OTHER OUTCOMES:
Software failure rate | 30seconds
The incidence of adverse events and serious adverse events | 30seconds

CONTACTS AND LOCATIONS:
Overall Officials: Guo Yutao, doctor, Principal Investigator — The First Medical Center of the Chinese PLA General Hospital & Medical School
Locations (2):
- China (2):
  - The First Medical Center of the Chinese PLA General Hospital & Medical School, Beijing
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou

IPD SHARING:
Plan to Share IPD: No